CLINICAL TRIAL: NCT01601886
Title: Delivery Room Practice Change Following the Initiation of the NICHD SUPPORT Trial
Status: Completed | Type: Observational
Sponsor: Luc Brion (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor-Investigator, Luc Brion, Professor of Pediatrics, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Other Study IDs: STU 092010-201; Velos 12121 (Other: University of Texas Southwestern)
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Preterm Birth
Keywords: Intubation, Intratracheal; Continuous Positive Airway Pressure; Historical Cohort Studies; Clinical Trial
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Before SUPPORT: 01/03-06/05
- During SUPPORT recruitment: 07/05-02/09
- After SUPPORT: 03/09-06/10

SUMMARY:
This study was designed to analyze whether initiation of the NICHD Neonatal Research Network SUPPORT trial was followed by a change in frequency of endotracheal intubation the delivery room in non-participants and whether these changes were associated with changes in management and outcomes.

The investigators hypothesized that the investigators would observe following the initiation of the SUPPORT trial a 33% reduction in the rate of intubation in the delivery room among non-participants preterm infants at Parkland Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

* All babies born at Parkland Memorial Hospital with gestational age at least 24 weeks and less than 35 weeks between 01/2003 and 06/2010

Exclusion Criteria:

* Infants receiving comfort care
* Those with major congenital anomalies
* Those enrolled in the SUPPORT trial

Ages: 24 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All babies born at Parkland Memorial Hospital with gestational age at least 24 weeks and less than 35 weeks between 01/2003 and 06/2010
Sampling Method: Non-Probability Sample
Enrollment: 3843 (Actual)
Dates: Start 2008-04; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Endotracheal intubation in the delivery room | In the delivery room (1 day)
  Frequency of endotracheal intubation in the delivery room

SECONDARY OUTCOMES:
Continuous positive airway pressure in the delivery room | In the delivery room (1 day)
  Frequency of continuous positive airway pressure in the delivery room
Endotracheal intubation in the first four hours after admission | First four hours after admission
  Frequency of endotracheal intubation in the first fours after admission to the neonatal intensive care unit
Endotracheal intubation until four hours after admission | Between birth and 4 hours after admission
  Frequency of endotracheal intubation between birth and four hours after admission in the neonatal intensive care unit
Admninistration of surfactant | Any time between birth and 2 days of age
  Frequency of admninistration of surfactant any time between birth and 2 days of age
Pneumothorax | Any time before discharge or transfer or 12 months of age (whichever comes first)
  Pneumothorax any time before discharge or transfer or 12 months of age (whichever comes first)
Bronchopulmonary dysplasia | 28 days
  Chronic changes on chest radiograph and oxygen requirement (fractional inspiratory concentration of oxygen greater than 0.21) for at least 28 days
Necrotizing enterocolitis | Any time before discharge or transfer or 12 months of age (whichever comes first)
  Necrotizing enterocolitis (at least stage II, modified Bell's classification) any time before discharge or transfer or 12 months of age (whichever comes first)
Duration of mechanical ventilation | Until discharge or transfer or 12 months of age (whichever comes first)
  Duration of invasive mechanical ventilation until discharge or transfer or or 12 months of age (whichever comes first)
Maximum oxygen concentration | Until discharge or transfer or 12 months of age (whichever comes first)
  Maximum inspiratory oxygen concentration until discharge or transfer or 12 months of age (whichever comes first)
Severe retinopathy of prematurity | Until discharge or transfer or 12 months of age (whichever comes first)
  Severe retinopathy of prematurity (at least stage III, international classification) until discharge or transfer or 12 months of age (whichever comes first)
Mortality | Until discharge or transfer or 12 months of age (whichever comes first)
  Mortality until discharge or transfer or 12 months of age (whichever comes first)
Severe brain lesion on imaging | Any time before discharge or transfer or 12 months of age (whichever comes first)
  Cystic periventricular leukomalacia or grade III or IV intraventricular/ periventricular hemorrhage detected by ultrasonogram any time before discharge or transfer or 12 months of age (whichever comes first)

CONTACTS AND LOCATIONS:
Overall Officials: Luc P Brion, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States